CLINICAL TRIAL: NCT05024318
Title: NeoAdjuvant Pembrolizumab and STEreotactic Radiotherapy Prior to Nephrectomy for Renal Cell Carcinoma: Investigating Induced Immune Context Changes
Brief Title: NeoAdjuvant Pembrolizumab and STEreotactic Radiotherapy Prior to Nephrectomy for Renal Cell Carcinoma
Acronym: NAPSTER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/007
Record Dates: First submitted 2021-03-29; First posted 2021-08-27 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Renal Cell Carcinoma, Clear Cell, Somatic
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; Nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SABR plus nephrectomy (Active Comparator): Stereotactic Ablative Radiotherapy (SABR) will be prescribed to a dose of 42Gy in 3 fractions. All radiotherapy treatment be completed within 3 weeks.Patients will undergo nephrectomy within 9-12 weeks after the first dose of treatment.
  Interventions: Radiation: Stereotactic Ablative Radiotherapy; Procedure: Nephrectomy
- Pembrolizumab followed by SABR after cycle 1 plus nephrectomy (Experimental): Pembrolizumab 200 mg (flat dose) will be administered as a 30 minute IV infusion every 21 days for 3 cycles. Patients will receive 1 cycle of pembolizumab prior to SABR followed by an additional 2 cycles of pembrolizumab (1 cycle is 21 days). Patients will undergo nephrectomy 9-12 weeks after commencement of treatment.
  Interventions: Drug: Pembrolizumab; Radiation: Stereotactic Ablative Radiotherapy; Procedure: Nephrectomy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg tobe administered as a 30 minute IV infusion every 21 days for 3 cycles
  Other Names: MK-3475
  Arms: Pembrolizumab followed by SABR after cycle 1 plus nephrectomy
Radiation: Stereotactic Ablative Radiotherapy — 42Gy delivered in 3 fractions
  Other Names: SABR
Procedure: Nephrectomy — Partial or total nephrectomy performed 9-12 weeks after first dose of Pembrolizumab
  Other Names: Surgical removal of a kidney

SUMMARY:
This is a prospective, open label, phase II, randomised, non-comparative clinical trial, evaluating changes in tumour-responsive T-cells following neoadjuvant stereotactic ablative body radiotherapy (SABR) with or without pembrolizumab, prior to nephrectomy, in patients with localised primary clear cell renal cell carcinoma (ccRCC).

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent
2. Male or female aged 18 years or older at written informed consent
3. Histologically or cytologically confirmed diagnosis of RCC with clear cell, rhabdoid or sarcomatoid components
4. Tumour stage T1B-T3, N0 or N1, M0 or low volume M1 planned for nephrectomy
5. Patients must have adequate bone marrow, hepatic and renal function documented within 28 days prior to randomisation:

   * White Blood Cell (WBC) ≥ 3 X 10^9/L
   * Absolute neutrophil count (ANC) ≥1.5 X 10^9/L
   * Platelets ≥ 100 X 10^9/L
   * Haemoglobin ≥ 100 g/L independent of transfusion
   * Serum Creatinine ≤1.5 X Upper Limit of Normal (ULN) or measured or calculated CrCl calculated as per institutional standard ≥ 30 ml/min. GFR can also be used in place of serum creatinine or CrCl.
   * Total bilirubin ≤1.5 X ULN except for patients with known Gilbert's Syndrome
   * Albumin > 30 g/L
   * AST and ALT ≤1.5 X ULN
   * INR or PT ≤1.5 X ULN unless patient is receiving anticoagulant therapy
6. ECOG performance status of 0 or 1
7. Women of child birth potential (WOCBP) must have a negative urine or serum pregnancy test within 72 hours prior to randomisation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
8. WOCBP should be willing to use two methods of birth control, or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilised or have not been free from menses for more than 1 year
9. Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
10. Patient agrees to the collection and use of their fresh tumour samples and peripheral blood for translational research
11. Patient is willing and able to comply with the protocol for the duration of the study including undergoing biopsies, treatment, and scheduled visits and examination

Exclusion Criteria:

1. Had prior treatment with any anti-PD-1, or anti-PD-L1, or PD-L2 agent or with an antibody targeting any other immune-regulatory receptors or mechanisms. Examples of such antibodies include antibodies against IDO, PD-L1, IL-2R, and GITR
2. Known or active inflammatory bowel disease involving colon and small bowels
3. Previous radiotherapy to the upper abdomen with radiation dose overlap to the involved kidney
4. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to randomisation
5. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy exceeding 10 mg daily dose of prednisone or equivalent or any other form of immunosuppressive therapy within 7 days prior to randomisation
6. Has an active autoimmune disease that has required systemic treatment in the last 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
7. Has a known additional malignancy that is progressing or has required active treatment in the last 2 years Note: Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ, such as breast cancer in situ, that has undergone potentially curative therapy are not excluded
8. Has known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to randomisation
9. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
10. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
11. Has an active infection requiring systemic therapy
12. Has a known history of HIV infection
13. Has known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive)or known active Hepatitis C (defined as HCV RNA [qualitative] is detected) infection
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
15. Has a known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
16. Has received a live virus vaccine within 30 days prior to randomisation. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed
17. Has had a prior solid organ transplant
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study drug.
19. Any contraindications for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
mPR post-SABR with or without pembrolizumab | At nephrectomy performed 9-12 weeks after first dose of pembrolizumab
  The mPR rate is defined as <10% residual tumour at post-nephrectomy specimens
CD8+ TRM in baseline biopsy and post-nephrectomy specimen, all measured as a continuous variable. | Baseline and at nephrectomy performed 9-12 weeks after first dose of pembrolizumab
  To describe changes in tumour-responsive T-cells, TRM CD8+ T-cells from baseline to post-nephrectomy in patients treated with SABR with or without pembrolizumab treatment followed by nephrectomy
TCF-1 + tumour infiltrating lymphocytes (TILs) in baseline biopsy and post-nephrectomy specimen, measured as a continuous variable | Baseline and at nephrectomy performed 9-12 weeks after first dose of pembrolizumab
  To describe changes in TCF-1+ T-cells from baseline to post-nephrectomy in patients treated with SABR with or without pembrolizumab treatment followed by nephrectomy

SECONDARY OUTCOMES:
Immune response cells in baseline biopsy and post-nephrectomy specimen | Baseline and at nephrectomy performed 9-12 weeks after first dose of pembrolizumab
  Change in immune response from baseline to post-nephrectomy
The tumour-responsive TRM cells inclusive of CD4+ and CD8+ compartments | 2 weeks prior to nephrectomy
  Percentage of tumour responsive T-cells (inclusive CD4/CD8) after neo-adjuvant treatment
Safety of SABR with or without pembrolizumab in the neo-adjuvant setting | 60 days post nephrectomy
  Adverse events, as measured by CTCAE v5.0
Change in immune response associated with mPR | Baseline and at nephrectomy performed 9-12 weeks after first dose of pembrolizumab
  Immune response cells in baseline biopsy and post-nephrectomy specimens
Change in PD-L1 and PD-L2 expression in tumour | Baseline and at nephrectomy performed 9-12 weeks after first dose of pembrolizumab
  PD-L1 and PD-L2 expression in baseline biopsy and post-nephrectomy specimens

OTHER OUTCOMES:
Radiological features including contrast enhancement consistent with mPR | 2 weeks prior to nephrectomy
  Post treatment radiological features including contrast enhancement
Radiological features including size reduction consistent with mPR | 2 weeks prior to nephrectomy
  Post treatment radiological features including size reduction
Radiological features including maximum tumour diameter consistent with mPR | 2 weeks prior to nephrectomy
  Post treatment radiological features including maximum tumour diameter
Radiological features including margins consistent with mPR | 2 weeks prior to nephrectomy
  Post treatment radiological features including margins
Baseline versus post-nephrectomy tissue for immune context changes | Baseline and at nephrectomy performed 9-12 weeks after first dose of pembrolizumab
  To investigate baseline versus post-nephrectomy tissue for immune context changes, using a broad panel of assays which will be further developed through the lifetime of the study
Baseline versus post-nephrectomy tissue immune network signalling | Baseline and at nephrectomy performed 9-12 weeks after first dose of pembrolizumab
  Baseline and post-nephrectomy immune network signalling , using a broad panel of assays which will be further developed through the lifetime of the study
Systemic immune cells in baseline and post-nephrectomy blood samples | Baseline and at nephrectomy performed 9-12 weeks after first dose of pembrolizumab
  To investigate changes in systemic immunity of patients with primary ccRCC treated with SABR with or without pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Shankar Siva, A/Prof, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (2):
- Australia (2):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No